CLINICAL TRIAL: NCT05788822
Title: A Single-center Randomized Controlled Trial on Mevalproic Acid Improving Oocyte Quality and Embryo Development in Elderly Infertile Patients
Brief Title: MVA to Improve the Pregnancy Outcome in Aged Infertility Women With Assisted Reproductive Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing University (Other)
Responsible Party: Principal Investigator, Li-jun Ding, reseaerch fellow, Nanjing University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SZ-MVA-1
Record Dates: First submitted 2023-03-13; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Infertility, Female; IVF; Reproductive Disorder; Oocyte
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MVA treated group (Experimental): Oocytes in this groups will be cultured with MVA
  Interventions: Dietary Supplement: Mevalproic acid
- Control group (No Intervention): Oocytes in this groups will be culture without MVA

INTERVENTIONS:
Dietary Supplement: Mevalproic acid — Methovalerate pathway is a metabolism of cholesterol and isoprenoid synthesized from acetyl coenzyme A Pathway, which plays a key role in human health and disease, is also necessary for human cells to maintain normal functions. There are a series of important metabolic intermediates in the mevalproate pathway, such as farnesyl diphosphate and incense Folyl vanillin diphosphates, which modify proteins through isoprene, play an important role in regulating cell function. In addition, the latest research shows that valproic acid, the key metabolic intermediate of valproic acid pathway, being the synthetic precursor of cholesterol and isoprene, it can activate insulin growth factor (IGF)1-R and mTOR signals and maintain cell function by mediating histone function
  Arms: MVA treated group

SUMMARY:
The goal of this clinical trial is to test MVA on improving pregnancy outcome in elderly infertile patients undergoing invitro fertilization (IVF). The main question it aims to answer is whether MVA could improve embryo haploid rate. Participants requested IVF are asked to randomly culture equal numbers of oocyte and embryo with or without MVA. Therefore, sibling oocytes were randomly divided into test group and control group.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants will write the informed contents. This study is a randomized controlled study co compare different treatment methods on the embryo development. Sibling eggs were randomly divided into test group and control group. Specific method of randomization: all the eggs of each subject were distributed into two dishes (dish 1 and dish 2). If the oocyte number is odd, put the extra oocyte into dish 1. Using statistical software, the two dishes were randomly treated as test group and control group. Thus, a random allocation table was generated and a separate random envelope was made for each subject. The random envelope is kept and distributed by the relevant personnel who are not involved in the screening and treatment of subjects and are authorized by the researcher. Each selected subject must open the random envelope. The subjects were subjected to routine ovulation promotion, and then the acquired oocytes and cumulus cell complexes (COCs) were obtained and fertilized in vitro. The test group oocytes were cultured with MVA, while the control oocytes were cultured without MVA. Thus, half of the eggs from each elderly infertile patient were treated with MVA.

ELIGIBILITY:
Inclusion Criteria:

1. 38 years ≤ age ≤ 42 years;
2. Number of IVF/ICSI cycles ≤ 2

Exclusion Criteria:

1. Egg donor cycle
2. Chromosome abnormality;
3. Adenomyosis, hysteromyoma, thin endometrium, endometriosis and other uterine diseases;
4. Patients with repeated implantation failure

Ages: 38 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Estimated)
Dates: Start 2022-10-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Embryo haploid rate | one month after oocyte retrival
  Preimplantation genetic testing (PGT) was used to test embryo haploid rate

CONTACTS AND LOCATIONS:
Overall Officials: Haixiang Sun, MD, Study Director — Center for Reproductive Medicine and Obstetrics and Gynecology, Drum Tower Hospital, Nanjing University Medical School
Locations (1):
- Reproductive Medicine Center, The affiliated Drum Towel Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No